CLINICAL TRIAL: NCT04601779
Title: INFANT HEALTH- Supporting Infants' Mental Health and Healthy Weight Development Through Community Health Nurses' Promoting Sensitive Parenting
Brief Title: INFANT HEALTH- Promoting Mental Health and Healthy Weight in Infancy Through Sensitive Parenting
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Danish Council for Independent Research (Other); The Novo Nordic Foundation (Other); University of Glasgow (Other); ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 95-110-21307
Record Dates: First submitted 2020-10-19; First posted 2020-10-26 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Infant Mental Health; Parenting; Parent-Child Relations
Keywords: Infant mental health; Regulatory problems; Developmental psychopathology; Video-feedback to Promote Positive Parenting, VIPP; Overeating in infancy; Infancy overweight

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cluster I (Other): Cluster I is randomized to start the VIPP-PUF intervention phase May 1, 2022
  Interventions: Behavioral: VIPP-PUF
- Cluster II (Other): Cluster II is randomized to start the VIPP-PUF intervention phase November 1, 2022
  Interventions: Behavioral: VIPP-PUF
- Cluster III (Other): Cluster IiI is randomized to start the VIPP-PUF intervention phase March 1, 2023
  Interventions: Behavioral: VIPP-PUF

INTERVENTIONS:
Behavioral: VIPP-PUF — The VIPP-PUF Intervention is developed as an add-on to the existing PUF-program to address infants with major cognitive and regulatory vulnerabilities identified at age 9-10 months and adapted to the settings of community health nurses. The intervention (VIPP-PUF) will be created from an evidence-based method, the Video-based Intervention to Promote Positive Parenting (VIPP), to comprise six therapeutic sessions delivered by the community health nurse during home visits over a three months period. The VIPP -PUF builds on teaching the health nurses to promote parents' sensitivity to meet infants' cognitive and regulatory vulnerabilities, while taking in account the particular needs of families of psycho-social disadvantage.

SUMMARY:
Mental health problems and overweight often co-occur, they have their origin in early childhood and new research evidence suggest a key role of cognitive, emotional and behavioral regulation in the early developmental trajectories and points to the benefits of intervention in infancy that builds on strategies of sensitive parenting.

The research group behind this project has developed the PUF program (PUF: In Danish: 'Psykisk Udvikling og Funktion') to target infants' mental health and development within the settings of community health nurses. Still, measures are lacking that address the infants most vulnerable regarding the development and progression of mental health problems and overweight.

In this project, we develop and test a new intensified intervention to address major cognitive and regulatory vulnerabilities identified at child age 9-10 months and adapted to the settings of community health nurses. The intervention is created as an add-on to the PUF-program, using an evidence-based method to promote sensitive parenting, the Video-based Intervention to Promote Positive Parenting (VIPP). The new intervention VIPP-PUF comprises six therapeutic sessions delivered by the community health nurse during home visits over a three months period. The intervention builds on teaching the health nurses to promote parents' sensitivity to meet the infants' cognitive and regulatory vulnerabilities, and it takes in account the needs of psycho-socially disadvantaged families.

The Infant Health project is conducted in sixteen municipalities across Denmark. We use the Intervention Mapping approach as the study frame and integrate the best practice of community health nurses. The efficacy of the VIPP-PUF intervention is examined in a randomized controlled step-wedge design, in which approximately 1.000 children are followed up to the age of 24 months.

The VIPP-PUF intervention is hypothesized to reduce mental health problems at ages 24 months among infants with high levels of cognitive and regulatory problems at age 9-10 months, (primary outcome). Also, it is hypothesized that among children with high levels of cognitive and regulatory vulnerabilities at age 9-10 months, adding the VIPP-PUF intervention to treatment as usual at age 9-10 months, will reduce infants' cognitive and regulatory problems; promote healthy weight development; reduce parents' experiences of stress; promote sensitive parenting and promote parents' feeling of competence and relatedness.

DETAILED DESCRIPTION:
BACKGROUND Childhood mental health problems and overweight are highly prevalent, and they have severe long-term prognoses regarding mental and physical health, social functioning, and premature death.

The majority of child mental health problems have their origin within the first years of living with increased risk in infants from families of psycho-social disadvantage, and in infants with perinatal adversities and cognitive and psycho-motor difficulties. Problems of eating, sleep, and emotional and behavioral regulation may predict mental health problems and disorders and persistent dysregulation trajectories are associated with emotional- and behavioral problems, eating problems and attention deficit hyperactivity disorder, ADHD. Early parent-child relations and the quality of parenting has a key position in the risk mechanisms.

The risk of overweight is highly increased in children, who are overweight in infancy. Psycho-social risk factors are similar to those of mental health problems, e.g families of psycho-social disadvantage with risk mechanisms including gene-environment interaction, maternal feeding pattern; and higher risk among obese parents to introduce high energy and fat foods very early and having impaired responses to the infant's hunger and satiety cues.

Mental health problems tend to precede the development of overweight in childhood. Potential mechanisms include cognitive vulnerability of inhibitory control/reward, sensitivity and sustained attention, leading to impulsive eating and difficulties in delaying gratification. Infants' problems of emotional regulation and problems of maintaining an affective homeostasis confronted with stress-full experiences may result in emotional eating characterized by pathways of physiological stress responses and reward, in which appetite and attraction to sweet and fatty foods is considered to develop through poor emotional regulation and lower inhibitory control.

Prevention of mental health problems and overweight has to start early and combine universal strategies and targeted interventions to reduce risk exposures, optimize parenting and promote child development and a healthy weight development. The combination of universal approaches and specific intervention to target the most vulnerable children is the most effective way to the reduce the population load of childhood mental health problems and overweight.

Strategies to optimize parenting of infants at risk of mental health problems and overweight have to build on measures that promote parent's sensitivity, understanding and careful handling of the child's regulatory, emotional or cognitive vulnerabilities.

Home-visiting programs that are embedded in the general child health surveillance have unique possibilities of reaching the entire infant population and integrate specified interventions to infants and parents of particular needs.

The general child health surveillance in Denmark includes scheduled home visits to all infant families offered by community child health nurses, CHNs. The CHNs measure the child's weight and overall health and development, and they give parents advice regarding the care of the infant. In about 20% of infant families, the CHNs extend their services to target particular problems and needs, e.g regarding problems of eating and sleep, or the parent-child relation. Until recently, however, no standardized measures have been available to specifically address infants at risk of mental health problems and overweight. We have previously explored the possibilities of prevention within the municipality child health surveillance and identified potential predictors and mediators of developmental psychopathology, and a window of opportunity regarding intervention towards infants' cognitive and regulatory vulnerabilities at child age 9-10 months. We have developed, validated and implemented a standardized measure to help the CHNs to identify mental health vulnerabilities. By this measure, the CHNs combines information from parents and her own observations during the home-visit to make a final conclusion about the child's development and functioning within eight areas of child mental health: sleep, feeding and eating, emotional regulation, motor development, attention and concentration, curiosity and interests; contact and communication and language development. Validation studies have shown that children who have three or more problems within these areas have a significantly increased risk of mental health problems. The PUF-program was developed as a basic approach to help CHNs to guide their actions to address the problems identified at ages 9-10 months within the existing service settings. Still, the PUF-program do not include specified intervention to infants with high level of cognitive, regulatory and emotional problems, leaving these children behind with an increased risk of developing mental health problems and overweight.

AIMS The study aims to develop and test an intervention to promote sensitive parenting of infants with mental health vulnerabilities identified by CHNs at age 9-10 months and to be feasible within the settings of the municipality child health surveillance. Parents' resources are a particularly important regarding interventions to target child mental health and healthy weight, and it is a specific aim of the study to address the needs of parents of psycho-social adversities and how the intervention works for the most vulnerable families. The overall aim is to examine the feasibility, fidelity, and the effectiveness of the intervention delivered to parents of infants with major cognitive, regulatory and emotional problems with child mental health and weight development at child ages 18 and 24 months as the primary outcome.

METHODS The development, implementation and evaluation of the intervention is guided by the Intervention Mapping approach, guides for development of complex interventions from the UK Medical Research Council and the RE-AIM-method.

The Infant Health Study includes four work-packages (WPs), the WP 1: Project planning and management; WP 2: Creating the intervention; WP 3: The efficacy study; WP 4 the process evaluation, including an evaluation of what works for the vulnerable families, and a Pilot study prior to WP3 and WP 4.

The study is anchored in the settings of CHNs in a collaboration of municipalities who join a validated clinical database and among those municipalities who have implemented the basic PUF-program one year prior to study start. These municipalities are overall representative of the Danish population regarding key background characteristics.

The study is located at the National Institute of Public Health; and study methods make use of the particular opportunities of epidemiological research in Denmark due to a civil registration system which follows all citizens are throughout life and the possibilities of valid tracking of children, parents and background information from Danish population registries.

DESIGN The stepped wedge cluster randomized design is chosen because it is more feasible to randomize at the municipality level as compared to the level of the individual child or CHN. For practical reasons, all municipalities cannot be trained at the same time but have to be split into three groups, and with the stepped wedge design, we utilize this and randomly allocate the 16 participating municipalities to the time at which their health nurses have been trained, and at which they start offering the intervention to families. Also, with the stepped wedge design, spill over is reduced by the randomization of clusters as compared to individual randomization, and interventions are introduced in a stepwise manner to all participating clusters (municipalities in this case) which encourages participation for those who would otherwise have been randomized to the control condition. Further, with the stepped wedge design control families are recruited in the early phases of the trial, which enhances the recruiting of a control group with the level of usual care offered at the beginning of the trial. In the control period no participants receive intervention and sequential random crossover to the intervention cannot be reversed.

According to the randomization of municipalities, all children assessed to have high levels of cognitive and regulatory problems at age 9-10 months will function as controls and receive care as usual from Step 0 until the municipalities initiate the intervention in Step 1- 3, respectively.

PROJECTPLANNING AND MANAGEMENT (WP 1) A participatory planning group of the principal investigators and the leading CHNs are part of the planning and management of the project. A well-established collaboration with the leading CHNs from the participating municipalities facilitates their function as primary municipality stakeholders in WP 2-4.

The information from our close collaboration with the CHNs is currently updated in WP 1, and taken into account when developing the intervention, and in the strategies necessary to ensure fidelity and deliver valid results for the efficacy trial.

PREPARING THE INTERVENTION (WP 2) The overall goal is to create an intervention to function as an add-on to the basic PUF-program within the municipality settings in order to promote sensitive parenting of infants with high levels of cognitive and regulatory problems.

Among measures to promote parenting of vulnerable infants, the Video-feedback Intervention to Promote Positive Parenting, VIPP takes a strong position in being effective in the reduction of child problems, also in families of psycho-social disadvantage, including maternal eating problems. Research in effective obesity prevention in early childhood is scarce, but the available evidence points to infancy dysregulation and parenting as potential targets.

Initially, a group of CHNs are educated in the original VIPP method to enable them to contribute to the adaptation of the VIPP into the novel combined VIPP-PUF intervention. Further, these CHNs participate in the pilot testing of the VIPP-PUF, and they function as co-trainers and supervisors of the next generation of CHNs educated in the VIPP-PUF during the project period.

RECRUITMENT All children in the population are offered home visits, and more than 85% attend at the home visits at child age 9-10 months. Parents of children who have three or more problems at the PUF assessment are informed about the study by the CHNs, and via written folders and information on the study home page. If the parents agree to participate, they are afterwards invited to participate by e-post or by letter. Parents make their final agreement for participation by answering the web-based questionnaires at the study website. Parents who have difficulties in completing the questionnaires are offered assistance from the CHN. All participating parents get a gift certificate of about 27 euro after answering the questionnaires.

In the control phase of the study, the CHNs deliver their service and care as usual. In the intervention phase, the CHN offers parents the VIPP-PUF-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Three or more PUF problems at the PUF

Exclusion Criteria:

* Severe mental or physical illness or handicap.
* Not Danish or English speaking parents

Ages: 9 Months to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 406 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-05-17 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Child mental health | child age 24 months
  The Strengths and Difficulties Questionnaire (SDQ) answered by parents is used at ages 24 months in order to use this very short (25-items) and feasible measure both at age 24 months and at the planned follow-up at older ages.
  SDQ is highly predictive of persistent child mental health problems and suitable for the prospective investigation of mental health from ages 24 months and onwards. SDQ has been validated for use in children down to the age of 2 years, and used in epidemiological research worldwide, also in Danish populations, with Danish norms being available.
Social and emotional development | Child age 24 months
  The Ages and Stages Questionnaire, Social-Emotional 2 (ASQ: SE2) (version for children aged 1 to 60 months) is used to measure the child's self regulation, compliance, communication and adaptive functioning. It comprises 19 to 33 items rated by parents and includes a box parents in which parents may check if the behavior is a concern for them. The ASQ:SE2 is well-validated and the most commonly used measure of young children's social and emotional development, internationally as well as in Denmark.

SECONDARY OUTCOMES:
Weight-for-length z-scores | child age 24 months
  Weight-for-length z-scores are calculated from weight and lengths measured by CHNs at home visits using transportable scales and height carts and guidelines on how to perform the measurements.
Parenting | Child age 24 months
  The Being a Mother (BaM13)
Parental Stress | Child age 24 months
  The Parental Stress Scale (PSS). The scale is rated from 1-5 and values are summarised to a total PSS with some scores coded in the reverse order when relevant, with low total PSS scores being a better outcome.
Family impairment | Child age 24 months
  The WHO-5 well-being index (WHO-5)
Sensitive parenting | Child age 24 months
  Sensitive parenting will be examined from observer-ratings of video-recording of parent-infant interaction using the Child Interaction Behavior (CIB) system to assess the parent-child relationship. The CIB system contains 22 parent behavior codes, 16 child behavior codes, and five dyadic codes which can be aggregated into the following composites: sensitivity, intrusiveness, limit setting, involvement, withdrawal, compliance, dyadic reciprocity, and dyadic negative states. The CIB system has been validated in normative as well as high-risk populations, and shows stability over time, predictive validity and adequate psychometric properties.
  Coders will be trained to optimize intercoder reliability; and regular meetings and checks will be organized to prevent coder drift.
Eating behaviour and sensitive parenting during meals | Child age 24 months
  Video-recordings of mealtimes are used to examine the child's eating behaviour, the parents feeding behaviour, and the parent-child interaction with regard to parental sensitivity, intrusiveness and limit setting, regarding the child' involvement, withdrawal and compliance and concerning the overall dyadic reciprocity during a meal.
Parental feeding questionnaire | Child ages 18 and 24 months
  the Preschooler Feeding Questionnaire (PFQ) and the Child Feeding Questionnaire (CFQ) will be used to assess parent's perception of their feeding practices.
Child eating questionnaire | Child age 24 months
  The Child Eating Behavior Questionnaire (CEBQ) will be used to measure parent's perceptions of their child's eating behavior.
Child development progress | Child age 24 months
  The Ages and Stages Questionnaire, Third Edition (ASQ-3) consists of the following subscales: communication, gross motor, fine motor, problem-solving, and personal-social.

OTHER OUTCOMES:
Social and emotional development | Child at age 18 months
  The Ages and Stages Questionnaire, Social-Emotional 2 (ASQ: SE2) (version for children aged 1 to 60 months) is used to measure the child's self-regulation, compliance, communication and adaptive functioning. It comprises 19 to 33 items rated by parents and includes a box parents in which parents may check if the behavior is a concern for them. The ASQ SE2 is well-validated and the most commonly used measure of young children's social and emotional development, internationally as well as in Denmark.
Parenting | Child at age 18 months
  The Being a Mother (BaM 13)
Parental Stress | Child at age 18 months
  The Parental Stress Scale (PSS). The scale is rated from 1-5 and values are summarised to a total PSS with some scores coded in the reverse order when relevant, with low total PSS scores being a better outcome.
Family impairment | Child at age 18 months
  The WHO-5 well-being index (WHO-5)
Sensitive parenting | Child age 18 months
  Sensitive parenting will be examined from observer-ratings of video-recording of parent-infant interaction using the Child Interaction Behavior (CIB) system to assess the parent-child relationship. The CIB system contains 22 parent behavior codes, 16 child behavior codes, and five dyadic codes which can be aggregated into the following composites: sensitivity, intrusiveness, limit setting, involvement, withdrawal, compliance, dyadic reciprocity, and dyadic negative states. The CIB system has been validated in normative as well as high-risk populations, and shows stability over time, predictive validity and adequate psychometric properties.
  Coders will be trained to intercoder reliability ICC > .65, Pearson's r > .70, and regular meetings and checks will be organized to prevent coder drift.
Eating behavior incl overeating | Child age 18 months
  Parents answers questions on eating behaviour as part of the CBCL version 1 ½ -5.
Regulatory problems | Child age 18 months
  The Child Behaviour Checklist (CBCL) version for children aged 1 ½ -5 years, which includes information on regulatory problems of eating, sleep, emotions, behavioural and cognitive functions.
Parenting | Child age 18 months
  The Mother and Baby Interaction Scale (MABISC). The scale is rated from 0-4 and values are summarised to a total MABISC with some scores coded in the reverse order when relevant, with low total MABISC scores being a better outcome.
Body composition (bioimpedance) | Child age 24 months
  Body composition will be measured using bioimpedance which is feasible for use for children aged 24 months at a home visit. We will measure bioimpedance using the Impedimed SFB7 device (Impedimed, Brisbane, Australia) among 50 recruited children to calculate fat mass (FM) and fat-free mass (FFM). Based on previous literature on young children, we will use reference values for body composition for children to identify excess adiposity.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Mette Skovgaard, MD DM SCI, Principal Investigator — Professor; Morten Hulvej Rod, PhD, Study Director — Head of the National Institut of Public Health
Locations (1):
- National Institute of Public Health, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lancet Global Mental Health Group; Chisholm D, Flisher AJ, Lund C, Patel V, Saxena S, Thornicroft G, Tomlinson M. Scale up services for mental disorders: a call for action. Lancet. 2007 Oct 6;370(9594):1241-52. doi: 10.1016/S0140-6736(07)61242-2. PMID 17804059
- [Background] Erskine HE, Moffitt TE, Copeland WE, Costello EJ, Ferrari AJ, Patton G, Degenhardt L, Vos T, Whiteford HA, Scott JG. A heavy burden on young minds: the global burden of mental and substance use disorders in children and youth. Psychol Med. 2015 May;45(7):1551-63. doi: 10.1017/S0033291714002888. Epub 2014 Dec 23. PMID 25534496
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Murray CJ, Lopez AD. Global mortality, disability, and the contribution of risk factors: Global Burden of Disease Study. Lancet. 1997 May 17;349(9063):1436-42. doi: 10.1016/S0140-6736(96)07495-8. PMID 9164317
- [Background] Patel V, Flisher AJ, Hetrick S, McGorry P. Mental health of young people: a global public-health challenge. Lancet. 2007 Apr 14;369(9569):1302-1313. doi: 10.1016/S0140-6736(07)60368-7. PMID 17434406
- [Background] Lobstein T, Baur L, Uauy R; IASO International Obesity TaskForce. Obesity in children and young people: a crisis in public health. Obes Rev. 2004 May;5 Suppl 1:4-104. doi: 10.1111/j.1467-789X.2004.00133.x. No abstract available. PMID 15096099
- [Background] Swanson JD, Wadhwa PM. Developmental origins of child mental health disorders. J Child Psychol Psychiatry. 2008 Oct;49(10):1009-19. doi: 10.1111/j.1469-7610.2008.02014.x. No abstract available. PMID 19017021
- [Background] Costello EJ, Foley DL, Angold A. 10-year research update review: the epidemiology of child and adolescent psychiatric disorders: II. Developmental epidemiology. J Am Acad Child Adolesc Psychiatry. 2006 Jan;45(1):8-25. doi: 10.1097/01.chi.0000184929.41423.c0. PMID 16327577
- [Background] Skovgaard AM. Mental health problems and psychopathology in infancy and early childhood. An epidemiological study. Dan Med Bull. 2010 Oct;57(10):B4193. PMID 21040689
- [Background] Johnson MH, Gliga T, Jones E, Charman T. Annual research review: Infant development, autism, and ADHD--early pathways to emerging disorders. J Child Psychol Psychiatry. 2015 Mar;56(3):228-47. doi: 10.1111/jcpp.12328. Epub 2014 Sep 30. PMID 25266278
- [Background] Skovgaard AM, Houmann T, Christiansen E, Landorph S, Jorgensen T; CCC 2000 Study Team; Olsen EM, Heering K, Kaas-Nielsen S, Samberg V, Lichtenberg A. The prevalence of mental health problems in children 1(1/2) years of age - the Copenhagen Child Cohort 2000. J Child Psychol Psychiatry. 2007 Jan;48(1):62-70. doi: 10.1111/j.1469-7610.2006.01659.x. PMID 17244271
- [Background] Zeanah CH, Boris NW, Larrieu JA. Infant development and developmental risk: a review of the past 10 years. J Am Acad Child Adolesc Psychiatry. 1997 Feb;36(2):165-78. doi: 10.1097/00004583-199702000-00007. PMID 9031569
- [Background] Elberling H, Linneberg A, Olsen EM, Houmann T, Rask CU, Goodman R, Skovgaard AM. Infancy predictors of hyperkinetic and pervasive developmental disorders at ages 5-7 years: results from the Copenhagen Child Cohort CCC2000. J Child Psychol Psychiatry. 2014 Dec;55(12):1328-35. doi: 10.1111/jcpp.12256. Epub 2014 May 30. PMID 24889385
- [Background] Costello EJ. Early Detection and Prevention of Mental Health Problems: Developmental Epidemiology and Systems of Support. J Clin Child Adolesc Psychol. 2016 Nov-Dec;45(6):710-717. doi: 10.1080/15374416.2016.1236728. Epub 2016 Nov 18. PMID 27858462
- [Background] Lemcke S, Parner ET, Bjerrum M, Thomsen PH, Lauritsen MB. Early development in children that are later diagnosed with disorders of attention and activity: a longitudinal study in the Danish National Birth Cohort. Eur Child Adolesc Psychiatry. 2016 Oct;25(10):1055-66. doi: 10.1007/s00787-016-0825-6. Epub 2016 Feb 9. PMID 26861952
- [Background] Koch SV, Andersson M, Hvelplund C, Skovgaard AM. Mental disorders in referred 0-3-year-old children: a population-based study of incidence, comorbidity and perinatal risk factors. Eur Child Adolesc Psychiatry. 2021 Aug;30(8):1251-1262. doi: 10.1007/s00787-020-01616-2. Epub 2020 Aug 20. PMID 32815033
- [Background] Jaspers M, de Winter AF, Buitelaar JK, Verhulst FC, Reijneveld SA, Hartman CA. Early childhood assessments of community pediatric professionals predict autism spectrum and attention deficit hyperactivity problems. J Abnorm Child Psychol. 2013 Jan;41(1):71-80. doi: 10.1007/s10802-012-9653-4. PMID 22688680
- [Background] Shephard E, Bedford R, Milosavljevic B, Gliga T, Jones EJH, Pickles A, Johnson MH, Charman T; BASIS Team. Early developmental pathways to childhood symptoms of attention-deficit hyperactivity disorder, anxiety and autism spectrum disorder. J Child Psychol Psychiatry. 2019 Sep;60(9):963-974. doi: 10.1111/jcpp.12947. Epub 2018 Jul 2. PMID 29963709
- [Background] Skovgaard AM, Olsen EM, Christiansen E, Houmann T, Landorph SL, Jorgensen T; CCC 2000 Study Group. Predictors (0-10 months) of psychopathology at age 11/2 years - a general population study in The Copenhagen Child Cohort CCC 2000. J Child Psychol Psychiatry. 2008 May;49(5):553-62. doi: 10.1111/j.1469-7610.2007.01860.x. Epub 2008 Mar 10. PMID 18341552
- [Background] Rutter M, Kim-Cohen J, Maughan B. Continuities and discontinuities in psychopathology between childhood and adult life. J Child Psychol Psychiatry. 2006 Mar-Apr;47(3-4):276-95. doi: 10.1111/j.1469-7610.2006.01614.x. PMID 16492260
- [Background] Hemmi MH, Wolke D, Schneider S. Associations between problems with crying, sleeping and/or feeding in infancy and long-term behavioural outcomes in childhood: a meta-analysis. Arch Dis Child. 2011 Jul;96(7):622-9. doi: 10.1136/adc.2010.191312. Epub 2011 Apr 20. PMID 21508059
- [Background] Lemcke S, Parner ET, Bjerrum M, Thomsen PH, Lauritsen MB. EARLY REGULATION IN CHILDREN WHO ARE LATER DIAGNOSED WITH AUTISM SPECTRUM DISORDER. A LONGITUDINAL STUDY WITHIN THE DANISH NATIONAL BIRTH COHORT. Infant Ment Health J. 2018 Mar;39(2):170-182. doi: 10.1002/imhj.21701. Epub 2018 Feb 27. PMID 29485729
- [Background] Breeman LD, Jaekel J, Baumann N, Bartmann P, Bauml JG, Avram M, Sorg C, Wolke D. Infant regulatory problems, parenting quality and childhood attention problems. Early Hum Dev. 2018 Sep;124:11-16. doi: 10.1016/j.earlhumdev.2018.07.009. Epub 2018 Aug 2. PMID 30077865
- [Background] Cook F, Giallo R, Hiscock H, Mensah F, Sanchez K, Reilly S. Infant Regulation and Child Mental Health Concerns: A Longitudinal Study. Pediatrics. 2019 Mar;143(3):e20180977. doi: 10.1542/peds.2018-0977. Epub 2019 Feb 8. PMID 30737245
- [Background] Hyde R, O'Callaghan MJ, Bor W, Williams GM, Najman JM. Long-term outcomes of infant behavioral dysregulation. Pediatrics. 2012 Nov;130(5):e1243-51. doi: 10.1542/peds.2010-3517. Epub 2012 Oct 1. PMID 23027170
- [Background] Winsper C, Wolke D. Infant and toddler crying, sleeping and feeding problems and trajectories of dysregulated behavior across childhood. J Abnorm Child Psychol. 2014;42(5):831-43. doi: 10.1007/s10802-013-9813-1. PMID 24122374
- [Background] Poustka L, Zohsel K, Blomeyer D, Jennen-Steinmetz C, Schmid B, Trautmann-Villalba P, Hohmann S, Becker K, Esser G, Schmidt MH, Brandeis D, Banaschewski T, Laucht M. Interacting effects of maternal responsiveness, infant regulatory problems and dopamine D4 receptor gene in the development of dysregulation during childhood: A longitudinal analysis. J Psychiatr Res. 2015 Nov;70:83-90. doi: 10.1016/j.jpsychires.2015.08.018. Epub 2015 Aug 29. PMID 26424426
- [Background] Boe T, Sivertsen B, Heiervang E, Goodman R, Lundervold AJ, Hysing M. Socioeconomic status and child mental health: the role of parental emotional well-being and parenting practices. J Abnorm Child Psychol. 2014;42(5):705-15. doi: 10.1007/s10802-013-9818-9. PMID 24150864
- [Background] Laucht M, Esser G, Baving L, Gerhold M, Hoesch I, Ihle W, Steigleider P, Stock B, Stoehr RM, Weindrich D, Schmidt MH. Behavioral sequelae of perinatal insults and early family adversity at 8 years of age. J Am Acad Child Adolesc Psychiatry. 2000 Oct;39(10):1229-37. doi: 10.1097/00004583-200010000-00009. PMID 11026176
- [Background] Lucassen N, Kok R, Bakermans-Kranenburg MJ, Van Ijzendoorn MH, Jaddoe VW, Hofman A, Verhulst FC, Lambregtse-Van den Berg MP, Tiemeier H. Executive functions in early childhood: the role of maternal and paternal parenting practices. Br J Dev Psychol. 2015 Nov;33(4):489-505. doi: 10.1111/bjdp.12112. Epub 2015 Sep 10. PMID 26359942
- [Background] Loman MM, Gunnar MR; Early Experience, Stress, and Neurobehavioral Development Center. Early experience and the development of stress reactivity and regulation in children. Neurosci Biobehav Rev. 2010 May;34(6):867-76. doi: 10.1016/j.neubiorev.2009.05.007. Epub 2009 May 27. PMID 19481109
- [Background] Ryan R, O'Farrelly C, Ramchandani P. Parenting and child mental health. London J Prim Care (Abingdon). 2017 Aug 10;9(6):86-94. doi: 10.1080/17571472.2017.1361630. eCollection 2017 Nov. PMID 29181091
- [Background] Peneau S, Rouchaud A, Rolland-Cachera MF, Arnault N, Hercberg S, Castetbon K. Body size and growth from birth to 2 years and risk of overweight at 7-9 years. Int J Pediatr Obes. 2011 Jun;6(2-2):e162-9. doi: 10.3109/17477166.2010.518241. Epub 2010 Oct 28. PMID 20979545
- [Background] Baird J, Fisher D, Lucas P, Kleijnen J, Roberts H, Law C. Being big or growing fast: systematic review of size and growth in infancy and later obesity. BMJ. 2005 Oct 22;331(7522):929. doi: 10.1136/bmj.38586.411273.E0. Epub 2005 Oct 14. PMID 16227306
- [Background] Ester WA, Jansen PW, Hoek HW, Verhulst FC, Jaddoe VW, Marques AH, Tiemeier H, Susser ES, Roza SJ. Fetal size and eating behaviour in childhood: a prospective cohort study. Int J Epidemiol. 2019 Feb 1;48(1):124-133. doi: 10.1093/ije/dyy256. PMID 30508111
- [Background] Monteiro PO, Victora CG. Rapid growth in infancy and childhood and obesity in later life--a systematic review. Obes Rev. 2005 May;6(2):143-54. doi: 10.1111/j.1467-789X.2005.00183.x. PMID 15836465
- [Background] Druet C, Stettler N, Sharp S, Simmons RK, Cooper C, Smith GD, Ekelund U, Levy-Marchal C, Jarvelin MR, Kuh D, Ong KK. Prediction of childhood obesity by infancy weight gain: an individual-level meta-analysis. Paediatr Perinat Epidemiol. 2012 Jan;26(1):19-26. doi: 10.1111/j.1365-3016.2011.01213.x. Epub 2011 Aug 1. PMID 22150704
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in body-mass index, underweight, overweight, and obesity from 1975 to 2016: a pooled analysis of 2416 population-based measurement studies in 128.9 million children, adolescents, and adults. Lancet. 2017 Dec 16;390(10113):2627-2642. doi: 10.1016/S0140-6736(17)32129-3. Epub 2017 Oct 10. PMID 29029897
- [Background] Schmidt Morgen C, Rokholm B, Sjoberg Brixval C, Schou Andersen C, Geisler Andersen L, Rasmussen M, Nybo Andersen AM, Due P, Sorensen TI. Trends in prevalence of overweight and obesity in danish infants, children and adolescents--are we still on a plateau? PLoS One. 2013 Jul 24;8(7):e69860. doi: 10.1371/journal.pone.0069860. Print 2013. PMID 23894553
- [Background] Bammann K, Peplies J, De Henauw S, Hunsberger M, Molnar D, Moreno LA, Tornaritis M, Veidebaum T, Ahrens W, Siani A; IDEFICS Consortium. Early life course risk factors for childhood obesity: the IDEFICS case-control study. PLoS One. 2014 Feb 13;9(2):e86914. doi: 10.1371/journal.pone.0086914. eCollection 2014. PMID 24551043
- [Background] Aris IM, Bernard JY, Chen LW, Tint MT, Pang WW, Soh SE, Saw SM, Shek LP, Godfrey KM, Gluckman PD, Chong YS, Yap F, Kramer MS, Lee YS. Modifiable risk factors in the first 1000 days for subsequent risk of childhood overweight in an Asian cohort: significance of parental overweight status. Int J Obes (Lond). 2018 Jan;42(1):44-51. doi: 10.1038/ijo.2017.178. Epub 2017 Jul 28. PMID 28751763
- [Background] Woo Baidal JA, Locks LM, Cheng ER, Blake-Lamb TL, Perkins ME, Taveras EM. Risk Factors for Childhood Obesity in the First 1,000 Days: A Systematic Review. Am J Prev Med. 2016 Jun;50(6):761-779. doi: 10.1016/j.amepre.2015.11.012. Epub 2016 Feb 22. PMID 26916261
- [Background] Morgen CS, Andersen PK, Mortensen LH, Howe LD, Rasmussen M, Due P, Sorensen TI, Andersen AN. Socioeconomic disparities in birth weight and body mass index during infancy through age 7 years: a study within the Danish National Birth Cohort. BMJ Open. 2017 Jan 20;7(1):e011781. doi: 10.1136/bmjopen-2016-011781. PMID 28110282
- [Background] Morgen CS, Angquist L, Baker JL, Andersen AMN, Michaelsen KF, Sorensen TIA. Prenatal risk factors influencing childhood BMI and overweight independent of birth weight and infancy BMI: a path analysis within the Danish National Birth Cohort. Int J Obes (Lond). 2018 Apr;42(4):594-602. doi: 10.1038/ijo.2017.217. Epub 2017 Sep 8. PMID 28883541
- [Background] Thompson AL. Intergenerational impact of maternal obesity and postnatal feeding practices on pediatric obesity. Nutr Rev. 2013 Oct;71 Suppl 1(0 1):S55-61. doi: 10.1111/nure.12054. PMID 24147925
- [Background] DiSantis KI, Hodges EA, Johnson SL, Fisher JO. The role of responsive feeding in overweight during infancy and toddlerhood: a systematic review. Int J Obes (Lond). 2011 Apr;35(4):480-92. doi: 10.1038/ijo.2011.3. Epub 2011 Mar 22. PMID 21427696
- [Background] Hurley KM, Cross MB, Hughes SO. A systematic review of responsive feeding and child obesity in high-income countries. J Nutr. 2011 Mar;141(3):495-501. doi: 10.3945/jn.110.130047. Epub 2011 Jan 26. PMID 21270360
- [Background] Shloim N, Edelson LR, Martin N, Hetherington MM. Parenting Styles, Feeding Styles, Feeding Practices, and Weight Status in 4-12 Year-Old Children: A Systematic Review of the Literature. Front Psychol. 2015 Dec 14;6:1849. doi: 10.3389/fpsyg.2015.01849. eCollection 2015. PMID 26696920
- [Background] Blake-Lamb TL, Locks LM, Perkins ME, Woo Baidal JA, Cheng ER, Taveras EM. Interventions for Childhood Obesity in the First 1,000 Days A Systematic Review. Am J Prev Med. 2016 Jun;50(6):780-789. doi: 10.1016/j.amepre.2015.11.010. Epub 2016 Feb 22. PMID 26916260
- [Background] Anderson SE, Keim SA. Parent-Child Interaction, Self-Regulation, and Obesity Prevention in Early Childhood. Curr Obes Rep. 2016 Jun;5(2):192-200. doi: 10.1007/s13679-016-0208-9. PMID 27037572
- [Background] Glaus J, Cui L, Hommer R, Merikangas KR. Association between mood disorders and BMI/overweight using a family study approach. J Affect Disord. 2019 Apr 1;248:131-138. doi: 10.1016/j.jad.2019.01.011. Epub 2019 Jan 15. PMID 30731280
- [Background] Korczak DJ, Lipman E, Morrison K, Szatmari P. Are children and adolescents with psychiatric illness at risk for increased future body weight? A systematic review. Dev Med Child Neurol. 2013 Nov;55(11):980-7. doi: 10.1111/dmcn.12168. Epub 2013 Jun 7. PMID 23742661
- [Background] Korczak DJ, Lipman E, Morrison K, Duku E, Szatmari P. Child and adolescent psychopathology predicts increased adult body mass index: results from a prospective community sample. J Dev Behav Pediatr. 2014 Feb-Mar;35(2):108-17. doi: 10.1097/DBP.0000000000000015. PMID 24343190
- [Background] Luppino FS, de Wit LM, Bouvy PF, Stijnen T, Cuijpers P, Penninx BW, Zitman FG. Overweight, obesity, and depression: a systematic review and meta-analysis of longitudinal studies. Arch Gen Psychiatry. 2010 Mar;67(3):220-9. doi: 10.1001/archgenpsychiatry.2010.2. PMID 20194822
- [Background] Roberts RE, Duong HT. Obese youths are not more likely to become depressed, but depressed youths are more likely to become obese. Psychol Med. 2013 Oct;43(10):2143-51. doi: 10.1017/S0033291712002991. Epub 2013 Jan 9. PMID 23298458
- [Background] Cortese S, Moreira-Maia CR, St Fleur D, Morcillo-Penalver C, Rohde LA, Faraone SV. Association Between ADHD and Obesity: A Systematic Review and Meta-Analysis. Am J Psychiatry. 2016 Jan;173(1):34-43. doi: 10.1176/appi.ajp.2015.15020266. Epub 2015 Aug 28. PMID 26315982
- [Background] Schmidt Petersen MN, Houmann TB, Olsen EM. [Overweight and eating disorders in patients with attention deficit hyperactivity disorder]. Ugeskr Laeger. 2018 Jul 9;180(28):V11170877. Danish. PMID 29984707
- [Background] Nigg JT, Johnstone JM, Musser ED, Long HG, Willoughby MT, Shannon J. Attention-deficit/hyperactivity disorder (ADHD) and being overweight/obesity: New data and meta-analysis. Clin Psychol Rev. 2016 Feb;43:67-79. doi: 10.1016/j.cpr.2015.11.005. Epub 2015 Dec 2. PMID 26780581
- [Background] Bergmeier H, Skouteris H, Horwood S, Hooley M, Richardson B. Associations between child temperament, maternal feeding practices and child body mass index during the preschool years: a systematic review of the literature. Obes Rev. 2014 Jan;15(1):9-18. doi: 10.1111/obr.12066. Epub 2013 Aug 19. PMID 23957249
- [Background] Byrne ME, LeMay-Russell S, Tanofsky-Kraff M. Loss-of-Control Eating and Obesity Among Children and Adolescents. Curr Obes Rep. 2019 Mar;8(1):33-42. doi: 10.1007/s13679-019-0327-1. PMID 30701372
- [Background] Graziano PA, Calkins SD, Keane SP. Toddler self-regulation skills predict risk for pediatric obesity. Int J Obes (Lond). 2010 Apr;34(4):633-41. doi: 10.1038/ijo.2009.288. Epub 2010 Jan 12. PMID 20065961
- [Background] Graziano PA, Kelleher R, Calkins SD, Keane SP, Brien MO. Predicting weight outcomes in preadolescence: the role of toddlers' self-regulation skills and the temperament dimension of pleasure. Int J Obes (Lond). 2013 Jul;37(7):937-42. doi: 10.1038/ijo.2012.165. Epub 2012 Oct 9. PMID 23044856
- [Background] Aparicio E, Canals J, Arija V, De Henauw S, Michels N. The role of emotion regulation in childhood obesity: implications for prevention and treatment. Nutr Res Rev. 2016 Jun;29(1):17-29. doi: 10.1017/S0954422415000153. PMID 27045966
- [Background] Power TG, Olivera YA, Hill RA, Beck AD, Hopwood V, Garcia KS, Ramos GG, Fisher JO, O'Connor TM, Hughes SO. Emotion regulation strategies and childhood obesity in high risk preschoolers. Appetite. 2016 Dec 1;107:623-627. doi: 10.1016/j.appet.2016.09.008. Epub 2016 Sep 13. PMID 27620645
- [Background] Hughes SO, Power TG, O'Connor TM, Orlet Fisher J. Executive functioning, emotion regulation, eating self-regulation, and weight status in low-income preschool children: how do they relate? Appetite. 2015 Jun;89:1-9. doi: 10.1016/j.appet.2015.01.009. Epub 2015 Jan 14. PMID 25596501
- [Background] Saltzman JA, Liechty JM, Bost KK, Fiese BH; STRONG Kids Program. Parent binge eating and restrictive feeding practices: Indirect effects of parent's responses to child's negative emotion. Eat Behav. 2016 Apr;21:150-4. doi: 10.1016/j.eatbeh.2016.02.001. Epub 2016 Feb 26. PMID 26966790
- [Background] Saltzman JA, Pineros-Leano M, Liechty JM, Bost KK, Fiese BH; STRONG Kids Team. Eating, feeding, and feeling: emotional responsiveness mediates longitudinal associations between maternal binge eating, feeding practices, and child weight. Int J Behav Nutr Phys Act. 2016 Aug 2;13:89. doi: 10.1186/s12966-016-0415-5. PMID 27484590
- [Background] Conti G, Heckman JJ. The developmental approach to child and adult health. Pediatrics. 2013 Apr;131 Suppl 2(Suppl 2):S133-41. doi: 10.1542/peds.2013-0252d. PMID 23547057
- [Background] Arango C, Diaz-Caneja CM, McGorry PD, Rapoport J, Sommer IE, Vorstman JA, McDaid D, Marin O, Serrano-Drozdowskyj E, Freedman R, Carpenter W. Preventive strategies for mental health. Lancet Psychiatry. 2018 Jul;5(7):591-604. doi: 10.1016/S2215-0366(18)30057-9. Epub 2018 May 15. PMID 29773478
- [Background] Reilly JJ, Martin A, Hughes AR. Early-Life Obesity Prevention: Critique of Intervention Trials During the First One Thousand Days. Curr Obes Rep. 2017 Jun;6(2):127-133. doi: 10.1007/s13679-017-0255-x. PMID 28434107
- [Background] Vitaro F, Tremblay R. Clarifying and Maximizing the Usefulness of Targeted Preventive Interventions. In: Rutter M, Bishop D, Pine D, Scott S, Stevenson J, Taylor E, et al., editors. Rutter's Child and Adolescent Psychiatry. 5 ed. Oxford: Blackwell Publishing; 2008. p. 971-87.
- [Background] Beckwith L. Prevention Science and Prevention Programs. In: Zeanah CH, editor. Handbook of Infant Mental Health. 2 ed. New York: The Guilford Press; 2000. p. 439-56.
- [Background] Groh AM, Fearon RMP, van IJzendoorn MH, Bakermans-Kranenburg MJ, Roisman GI. Attachment in the Early Life Course: Meta-Analytic Evidence for Its Role in Socioemotional Development. Child Development Perspectives. 2017;11(1):70-6.
- [Background] Zeanah PD, Gleason MM. Infant Mental Health in Primary Health Care. In: Zeanah CH, editor. Handbook of Infant Mental Health. 3 ed. New York: The Guilford Press; 2009. p. 549-63.
- [Background] Huffman LC, Nichols M. Early Detection of Young Children's Mental Health Problems in Primary Care Settings. In: DelCarmen-Wiggins R, Carter A, editors. Handbook of Infant, Toddler, and Preschool Mental Health Assessment. New York: Oxford University Press, Inc.; 2004. p. 467-90.
- [Background] Smith JD, St George SM, Prado G. Family-Centered Positive Behavior Support Interventions in Early Childhood To Prevent Obesity. Child Dev. 2017 Mar;88(2):427-435. doi: 10.1111/cdev.12738. Epub 2017 Feb 13. PMID 28195411
- [Background] Askie L, Martin A, Espinoza D, Campbell K, Daniels LA, Hesketh K, et al. What does the EPOCH (early prevention of obesity in childhood) prospective meta-analysis tell us about early life obesity prevention? Obesity Research & Clinical Practice. 2014;14:184.
- [Background] Redsell SA, Edmonds B, Swift JA, Siriwardena AN, Weng S, Nathan D, Glazebrook C. Systematic review of randomised controlled trials of interventions that aim to reduce the risk, either directly or indirectly, of overweight and obesity in infancy and early childhood. Matern Child Nutr. 2016 Jan;12(1):24-38. doi: 10.1111/mcn.12184. Epub 2015 Apr 20. PMID 25894857
- [Background] Wen LM, Baur LA, Rissel C, Wardle K, Alperstein G, Simpson JM. Early intervention of multiple home visits to prevent childhood obesity in a disadvantaged population: a home-based randomised controlled trial (Healthy Beginnings Trial). BMC Public Health. 2007 May 10;7:76. doi: 10.1186/1471-2458-7-76. PMID 17490492
- [Background] Yavuz HM, van Ijzendoorn MH, Mesman J, van der Veek S. Interventions aimed at reducing obesity in early childhood: a meta-analysis of programs that involve parents. J Child Psychol Psychiatry. 2015 Jun;56(6):677-92. doi: 10.1111/jcpp.12330. Epub 2014 Oct 8. PMID 25292319
- [Background] Asmussen K, Feinstein L, Martin J, Chowdry H. Foundations for life: What works to support parent child interaction in the early years. London: Early Intervention Foundation. 2016.
- [Background] Skovgaard AM, Olsen EM, Houmann T, Christiansen E, Samberg V, Lichtenberg A, Jorgensen T. The Copenhagen County child cohort: design of a longitudinal study of child mental health. Scand J Public Health. 2005;33(3):197-202. doi: 10.1080/14034940510005662. PMID 16040460
- [Background] Skovgaard AM, Wilms L, Johansen A, Ammitzboll J, Holstein BE, Olsen EM. [Standardised measuring the health of infants and toddlers in community health services]. Ugeskr Laeger. 2018 Aug 20;180(34):V12170960. Danish. PMID 30152319
- [Background] Olsen EM, Petersen J, Skovgaard AM, Thomsen BL, Jorgensen T, Weile B. The growth pattern of 0-1-year-old Danish children, when screened by public health nurses--the Copenhagen County Child Cohort 2000. Ann Hum Biol. 2005 May-Jun;32(3):297-315. doi: 10.1080/03014460500068360. PMID 16099775
- [Background] Skovgaard AM, Houmann T, Christiansen E, Olsen EM, Landorph SL, Lichtenberg A, Jorgensen T. Can a general health surveillance between birth and 10 months identify children with mental disorder at 1(1/2) year? A case-control study nested in cohort CCC 2000. Eur Child Adolesc Psychiatry. 2008 Aug;17(5):290-8. doi: 10.1007/s00787-007-0666-4. Epub 2008 Feb 26. PMID 18301939
- [Background] Ammitzboll J, Holstein BE, Wilms L, Andersen A, Skovgaard AM. A new measure for infant mental health screening: development and initial validation. BMC Pediatr. 2016 Dec 1;16(1):197. doi: 10.1186/s12887-016-0744-1. PMID 27905887
- [Background] Ammitzboll J, Thygesen LC, Holstein BE, Andersen A, Skovgaard AM. Predictive validity of a service-setting-based measure to identify infancy mental health problems: a population-based cohort study. Eur Child Adolesc Psychiatry. 2018 Jun;27(6):711-723. doi: 10.1007/s00787-017-1069-9. Epub 2017 Oct 20. PMID 29052014
- [Background] Ammitzboll J, Skovgaard AM, Holstein BE, Andersen A, Kreiner S, Nielsen T. Construct validity of a service-setting based measure to identify mental health problems in infancy. PLoS One. 2019 Mar 28;14(3):e0214112. doi: 10.1371/journal.pone.0214112. eCollection 2019. PMID 30921359
- [Background] Bartholomew L, Parcel G, Kok G, Gottlieb N, Fernández M. Planning Health Promotion Programs - An intervention mapping approach. 3 ed. San Francisco: Jossey-Bass; 2011.
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Harden SM, Smith ML, Ory MG, Smith-Ray RL, Estabrooks PA, Glasgow RE. RE-AIM in Clinical, Community, and Corporate Settings: Perspectives, Strategies, and Recommendations to Enhance Public Health Impact. Front Public Health. 2018 Mar 22;6:71. doi: 10.3389/fpubh.2018.00071. eCollection 2018. PMID 29623270
- [Background] Thygesen LC, Ersboll AK. When the entire population is the sample: strengths and limitations in register-based epidemiology. Eur J Epidemiol. 2014 Aug;29(8):551-8. doi: 10.1007/s10654-013-9873-0. Epub 2014 Jan 10. PMID 24407880
- [Background] Schmidt M, Pedersen L, Sorensen HT. The Danish Civil Registration System as a tool in epidemiology. Eur J Epidemiol. 2014 Aug;29(8):541-9. doi: 10.1007/s10654-014-9930-3. Epub 2014 Jun 26. PMID 24965263
- [Background] Statistics Denmark. IDA - an Integrated Database for labour market research. Main report. Copenhagen: Statistics Denmark; 1991.
- [Background] Handley MA, Schillinger D, Shiboski S. Quasi-experimental designs in practice-based research settings: design and implementation considerations. J Am Board Fam Med. 2011 Sep-Oct;24(5):589-96. doi: 10.3122/jabfm.2011.05.110067. PMID 21900443
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Background] Woertman W, de Hoop E, Moerbeek M, Zuidema SU, Gerritsen DL, Teerenstra S. Stepped wedge designs could reduce the required sample size in cluster randomized trials. J Clin Epidemiol. 2013 Jul;66(7):752-8. doi: 10.1016/j.jclinepi.2013.01.009. Epub 2013 Mar 22. PMID 23523551
- [Background] Hemming K, Lilford R, Girling AJ. Stepped-wedge cluster randomised controlled trials: a generic framework including parallel and multiple-level designs. Stat Med. 2015 Jan 30;34(2):181-96. doi: 10.1002/sim.6325. Epub 2014 Oct 24. PMID 25346484
- [Background] Bayer J, Hiscock H, Scalzo K, Mathers M, McDonald M, Morris A, Birdseye J, Wake M. Systematic review of preventive interventions for children's mental health: what would work in Australian contexts? Aust N Z J Psychiatry. 2009 Aug;43(8):695-710. doi: 10.1080/00048670903001893. PMID 19629791
- [Background] Barlow J, Bergman H, Kornor H, Wei Y, Bennett C. Group-based parent training programmes for improving emotional and behavioural adjustment in young children. Cochrane Database Syst Rev. 2016 Aug 1;2016(8):CD003680. doi: 10.1002/14651858.CD003680.pub3. PMID 27478983
- [Background] Juffer F, Bakermans-Kranenburg MJ. Working with Video-feedback Intervention to promote Positive Parenting and Sensitive Discipline (VIPP-SD): A case study. J Clin Psychol. 2018 Aug;74(8):1346-1357. doi: 10.1002/jclp.22645. Epub 2018 May 21. PMID 29781521
- [Background] Bakermans-Kranenburg MJ, van IJzendoorn MH, Juffer F. Less is more: meta-analyses of sensitivity and attachment interventions in early childhood. Psychol Bull. 2003 Mar;129(2):195-215. doi: 10.1037/0033-2909.129.2.195. PMID 12696839
- [Background] Stein A, Woolley H, Senior R, Hertzmann L, Lovel M, Lee J, Cooper S, Wheatcroft R, Challacombe F, Patel P, Nicol-Harper R, Menzes P, Schmidt A, Juszczak E, Fairburn CG. Treating disturbances in the relationship between mothers with bulimic eating disorders and their infants: a randomized, controlled trial of video feedback. Am J Psychiatry. 2006 May;163(5):899-906. doi: 10.1176/ajp.2006.163.5.899. PMID 16648333
- [Background] Woolley H, Hertzmann L, Stein A. Video-feedback intervention with mothers with postnatal eating disorders and their infants. In: Juffer F, Bakermans-Kranenburg MJ, Van Ijzendoorn MH, editors. Promoting positive parenting: An Attachment-Based Intervention. New York: Taylor & Francis Group; 2008. p. 111-38.
- [Background] Matthey S. Assessing the experience of motherhood: the Being a Mother Scale (BaM-13). J Affect Disord. 2011 Jan;128(1-2):142-52. doi: 10.1016/j.jad.2010.06.032. Epub 2010 Jul 22. PMID 20655114
- [Background] Berry JO, Jones WH. The Parental Stress Scale: Initial psychometric evidence. Journal of Social and Personal Relationships. 1995;12(3):463-72.
- [Background] Pontoppidan M, Nielsen T, Kristensen IH. Psychometric properties of the Danish Parental Stress Scale: Rasch analysis in a sample of mothers with infants. PLoS One. 2018 Nov 7;13(11):e0205662. doi: 10.1371/journal.pone.0205662. eCollection 2018. PMID 30403692
- [Background] Bech P. Measuring the Dimension of Psychological General Well-Being by the Who-5. Quality of Life Newsletter. 2004;32:16.
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Achenbach TM, Rescorla LA. Manual for the ACEBA School-Age Forms & Profiles. Burlington: University of Vermont, Research Center for Children, Youth and Families; 2000
- [Background] Goodman R, Ford T, Simmons H, Gatward R, Meltzer H. Using the Strengths and Difficulties Questionnaire (SDQ) to screen for child psychiatric disorders in a community sample. Br J Psychiatry. 2000 Dec;177:534-9. doi: 10.1192/bjp.177.6.534. PMID 11102329
- [Background] Goodman A, Goodman R. Strengths and difficulties questionnaire as a dimensional measure of child mental health. J Am Acad Child Adolesc Psychiatry. 2009 Apr;48(4):400-403. doi: 10.1097/CHI.0b013e3181985068. PMID 19242383
- [Background] Croft S, Stride C, Maughan B, Rowe R. Validity of the strengths and difficulties questionnaire in preschool-aged children. Pediatrics. 2015 May;135(5):e1210-9. doi: 10.1542/peds.2014-2920. Epub 2015 Apr 6. PMID 25847804
- [Background] D'Souza S, Waldie KE, Peterson ER, Underwood L, Morton SM. Psychometric Properties and Normative Data for the Preschool Strengths and Difficulties Questionnaire in Two-Year-Old Children. J Abnorm Child Psychol. 2017 Feb;45(2):345-357. doi: 10.1007/s10802-016-0176-2. PMID 27334707
- [Background] Niclasen J, Teasdale TW, Andersen AM, Skovgaard AM, Elberling H, Obel C. Psychometric properties of the Danish Strength and Difficulties Questionnaire: the SDQ assessed for more than 70,000 raters in four different cohorts. PLoS One. 2012;7(2):e32025. doi: 10.1371/journal.pone.0032025. Epub 2012 Feb 27. PMID 22384129
- [Background] Squires J, Bricker D, Twombly E. ASQ:SE-2 user's guide: Ages & Stages Questionnaires social-emotional. Paul H. Brookes Publishing Co. Inc; 2015.
- [Background] Pontoppidan M, Klest SK, Sandoy TM. The Incredible Years Parents and Babies Program: A Pilot Randomized Controlled Trial. PLoS One. 2016 Dec 14;11(12):e0167592. doi: 10.1371/journal.pone.0167592. eCollection 2016. PMID 27974857
- [Background] Trillingsgaard T, Maimburg RD, Simonsen M. The Family Startup Program: study protocol for a randomized controlled trial of a universal group-based parenting support program. BMC Public Health. 2015 Apr 21;15:409. doi: 10.1186/s12889-015-1732-3. PMID 25895494
- [Background] Vaever MS, Smith-Nielsen J, Lange T. Copenhagen infant mental health project: study protocol for a randomized controlled trial comparing circle of security -parenting and care as usual as interventions targeting infant mental health risks. BMC Psychol. 2016 Nov 22;4(1):57. doi: 10.1186/s40359-016-0166-8. PMID 27876079
- [Background] Feldman R. Parenting behavior as the environment where children grow. In: Mayes L, Lewis M, editors. The Cambridge Handbook of Environment in Human Development. New York: Cambridge University Press; 2012. p. 535-67.
- [Background] Whitcomb SA, Merrell KW. Behavioral, Social, and Emotional Assessment of Children and Adolescents. 4. ed. New York: Taylor & Francis; 2013.
- [Background] Feldman R. The relational basis of adolescent adjustment: trajectories of mother-child interactive behaviors from infancy to adolescence shape adolescents' adaptation. Attach Hum Dev. 2010 Jan;12(1-2):173-92. doi: 10.1080/14616730903282472. PMID 20390528
- [Background] Feldman R, Bamberger E, Kanat-Maymon Y. Parent-specific reciprocity from infancy to adolescence shapes children's social competence and dialogical skills. Attach Hum Dev. 2013;15(4):407-23. doi: 10.1080/14616734.2013.782650. Epub 2013 Apr 2. PMID 23544455
- [Background] Feldman R, Eidelman AI. Neonatal state organization, neuromaturation, mother-infant interaction, and cognitive development in small-for-gestational-age premature infants. Pediatrics. 2006 Sep;118(3):e869-78. doi: 10.1542/peds.2005-2040. Epub 2006 Jul 31. PMID 16880249
- [Background] Feldman R, Weller A, Sirota L, Eidelman AI. Testing a family intervention hypothesis: the contribution of mother-infant skin-to-skin contact (kangaroo care) to family interaction, proximity, and touch. J Fam Psychol. 2003 Mar;17(1):94-107. PMID 12666466
- [Background] Hackney M, Braithwaite S, Radcliff G. Postnatal depression: the development of a self-report scale. Health Visitor. 1996;69:103-4.
- [Background] Hoivik MS, Burkeland NA, Linaker OM, Berg-Nielsen TS. The Mother and Baby Interaction Scale: a valid broadband instrument for efficient screening of postpartum interaction? A preliminary validation in a Norwegian community sample. Scand J Caring Sci. 2013 Sep;27(3):733-9. doi: 10.1111/j.1471-6712.2012.01060.x. Epub 2012 Aug 14. PMID 22892011
- [Derived] Skovgaard AM, Bakermans-Kranenburg M, Pontoppidan M, Tjornhoj-Thomsen T, Madsen KR, Voss I, Wehner SK, Pedersen TP, Finseth L, Taylor RS, Tolstrup JS, Ammitzboll J. The Infant Health Study - Promoting mental health and healthy weight through sensitive parenting to infants with cognitive, emotional, and regulatory vulnerabilities: protocol for a stepped-wedge cluster-randomized trial and a process evaluation within municipality settings. BMC Public Health. 2022 Jan 28;22(1):194. doi: 10.1186/s12889-022-12551-z. PMID 35090411
- See also: World Health Organization. Childhood overweight and obesity 2016 — http://www.who.int/dietphysicalactivity/childhood/en/
- See also: SDQ Danish home page — http://www.sdq.dk

DOCUMENTS (1):
  • Study Protocol (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT04601779/Prot_002.pdf